CLINICAL TRIAL: NCT03730818
Title: Effects of Water-based Versus Land-based Exercise on Cancer-related Fatigue and Functional Capacity in Breast Cancer Survivors
Brief Title: Water-based Versus Land-based Exercise for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital del Mar (Other); Centre Esportiu Claror Marítim (Unknown)
Responsible Party: Principal Investigator, Raquel Sebio, Principal Investigator, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AQUAFIT-2018
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Exercise Therapy; Aquatic Therapy; Health-Related Quality of Life; Cancer-related Fatigue; Exercise Tolerance; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is an assessor-blind study. Physiotherapist in charge of performing the baseline and post-intervention assessment will be blinded to participants allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water-based Exercise Group (Experimental): The Water-based Exercise Group will compromise participants attending a 2 weekly exercise intervention each session lasting 1 hour for 12 weeks.
  Each session will consist of:
  * 10 minutes of warm-up: general mobilisation, walking, active stretching
  * 40 minutes of global training: 20 minutes of endurance exercise and 20 minutes of resistance exercises targeting large main muscle groups involved in daily life activities (squats, lateral hip abduction, row, etc.) using body weight and elastic bands
  * 10 minutes of cooling down: stretching, breathing exercises and relaxation Intensity will be monitored with the modified Borg Scale to maintain a 5 - 6 level of exertion during the first 5 weeks and progressively increase to a 6 - 7 level for the following weeks.
  Interventions: Other: Water-based Exercise Group
- Land-based Exercise Group (Active Comparator): The land-based exercise group will attend as well 2 weekly sessions lasting 1 hour each for 12 weeks.
  Each session will consist of the same structure as the Water-based Exercise Group including:
  * 10 minutes warm up
  * 40 minutes of global training (20 minutes of endurance exercise and 20 minutes of resistance training)
  * 10 minutes cool down. The exercises will be adapted from the water-based exercise group to match the requirements on the water-based exercise group. Intensity will be monitored with the Perceived Rate of Exertion Scale (modified Borg Scale, Borg 1982) to maintain a 5 - 6 level of exertion during the first 5 weeks and progressively increase to a 6 - 7 level for the following weeks.
  Interventions: Other: Land-based Exercise Group

INTERVENTIONS:
Other: Water-based Exercise Group — The intervention consist will of a water-based exercise protocol
  Arms: Water-based Exercise Group
Other: Land-based Exercise Group — The intervention will consist of a land-based exercise protocol
  Arms: Land-based Exercise Group

SUMMARY:
Physical activity and exercise have demonstrated to be an integral part of the cancer-continuum care. Despite strong evidence suggesting that both endurance and strength training should be encourage in cancer patients, there is still controversy regarding exercise dosage, frequency, volume and optimal environment of delivery. In this randomised controlled trial we aim to compare water-based versus land-based exercise in breast cancer survivors to decrease cancer-related fatigue (CRF), improve Health-Related Quality of Life (HRQoL), exercise tolerance, muscle strength and physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer patients post cancer treatment (at least for 6 months)
* Cancer-free at the time of recruitment
* Signed informed consent
* Living in the metropolitan area of Barcelona

Exclusion Criteria:

* Fear of water
* Receiving cancer therapy at the time of recruitment
* Not willing to participate/Refuse to sign informed consent
* Physical of cognitive impairments precluding the patient to perform the exercises

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in Cancer-related Fatigue | Cancer-related fatigue from baseline throughout the study period (24 weeks)
  Cancer-related fatigue as measure with the specific subscale found in the EORTC QLQ C30 questionnaire specifically designed for a cancer population

SECONDARY OUTCOMES:
Change in Exercise Functional Capacity | Exercise functional capacity from baseline throughout the study period (24 weeks)
  6 Minute Walk Test performed accordingly to international guidelines
Change in Physical Activity levels | Physical activity levels from baseline throughout the study period (24 weeks)
  Physical Activity in METS-hour/week and minutes/week assessed with a triaxial accelerometer (Actigraph wgt3x-bt)
Change in Upper Body Strength | Upper body strength from baseline throughout the study period (24 weeks)
  Upper body muscle strength measured with a hand-held dynamometer and a handgrip test
Change in Lower Body Strength | Lower body strength from baseline throughout the study period (24 weeks)
  Lower body muscle strength measured with a hand-held dynamometer (leg extension) and the sit-to-stand test
Change in Health-Related Quality of Life | Health-related quality of life from baseline throughout the study period (24 weeks)
  HRQoL measured with the EORTC QLQ C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Claror - Fundació Marítim, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No